CLINICAL TRIAL: NCT06880887
Title: The Acute Effects of Vagus Nerve Stimulation on the Autonomic Nervous System and Spasticity in Children with Spastic Cerebral Palsy
Brief Title: Nervus Vagus Stimulation and Cerebral Palsy
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, gulay karacaoglu, Assitant prof., Istanbul Medipol University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-526
Record Dates: First submitted 2025-03-10; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Palsy, Spastic
Keywords: autonomic nervus system activity; nervus vagus stimulation; asworth scala
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Since the acute effect of transcutaneous auricular vagus nerve stimulation on spasticity in children with spastic cerebral palsy was to be measured, all participants received the auricular vagus nerve stimulation intervention once.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- nervus vagus stimulation (Other): Since the acute effect of transcutaneous auricular vagus nerve stimulation on spasticity in children with spastic cerebral palsy was to be measured, all participants received the auricular vagus nerve stimulation intervention once.
  Interventions: Other: nervus vagus stimulation

INTERVENTIONS:
Other: nervus vagus stimulation — Vagus stimulation was applied bilaterally through the ear in a transcutaneous manner. transcutaneous auricular VNS (taVNS) was performed using the Vagustim device. The stimulation was applied for 20 minutes with a pulse width of 300 microseconds, a frequency of 10 Hz, and in a biphasic manner. The electrodes were placed on the concha and tragus parts of the ear, and the current was increased until the participant could feel it.

SUMMARY:
When the literature is reviewed, it is difficult to find direct research on the effects of auricular vagus nerve stimulation (aVNS) on the autonomic nervous system and spasticity in children with spastic cerebral palsy. However, there is a substantial body of literature on the potential of vagus nerve stimulation (VNS) to modulate autonomic functions.

The aim of this study is to investigate the potential effects of vagus nerve stimulation, which is known to influence the autonomic nervous system, in individuals with spastic cerebral palsy and to explore its contributions to spasticity.

DETAILED DESCRIPTION:
Individuals aged 2-15 years who applied to the Physical Medicine and Rehabilitation Department of Bursa VM Medical Park Hospital and were diagnosed with cerebral palsy (CP) by a physical medicine and rehabilitation physician or neurologist will be included in the study. A total of 20 participants were included in the study, and the necessary measurements were taken before and after the intervention.

The demographic characteristics of participants who meet the inclusion criteria will be recorded. After collecting sociodemographic characteristics, the following assessment methods will be applied, and the results will be recorded in the pre- and post-intervention evaluation form.

Evaluation After collecting the sociodemographic information of the included individuals, their Gross Motor Function Classification System (GMFCS) levels will be assessed and recorded. GMFCS is a scale that evaluates and classifies the gross motor skills of children with CP. It determines the walking abilities and levels of independence in physical activities of the children.

The 5 levels of GMFCS are defined as follows:

Level I (High Functional Level): Children at this level can walk and show limited success in complex movements such as running. They can usually climb stairs and use motor skills independently.

Level II (Moderate-High Functional Level): Children may have difficulty walking or running long distances but can walk. They may need support when climbing stairs and may require assistance to overcome obstacles.

Level III (Moderate Functional Level): Children at this level can walk but may need assistive devices (e.g., walkers) for shorter distances. They may require support when climbing stairs and assistance to overcome obstacles.

Level IV (Low Functional Level): Children can move independently only to a limited extent. Assistance may be required for walking or mobility, and they often use wheelchairs.

Level V (Very Low Functional Level): Children at this level are completely dependent and have difficulty performing any gross motor skills. They often require full support and have limited mobility.

Sociodemographic Information The names, ages, heights, weights, body mass indices (BMI), and diagnosis times of the individuals with CP included in the study will be recorded.

Spasticity Assessment:

The Modified Ashworth Scale (MAS) is a widely used tool to assess spasticity, measuring muscle tone associated with neurological conditions such as cerebral palsy, stroke, and spinal cord injuries. Spasticity can cause abnormal muscle contractions and movement limitations. MAS, which will be used in our study, determines the degree of muscle tone, allowing for a more objective evaluation of treatment and intervention needs.

The Modified Ashworth Scale evaluates the level of resistance exhibited by the muscle and typically detects the inability of the muscle to relax during joint movements. This scale measures the severity of spasticity on a grading system from 0 to 4:

0: No spasticity.

1. Slight increase in muscle tone, but no significant resistance during movement. 1+: Increased muscle tone with slight resistance during movement.
2. More noticeable increase in muscle tone, but joint movement is possible.
3. Significant increase in muscle tone, making joint movement difficult.
4. Muscle tone is so high that joint movement is not possible. MAS provides a simple, quick, and reliable method for monitoring spasticity. Its validity and reliability in different clinical conditions and treatment processes have been widely studied in the literature. For example, Bohannon and Smith (1987) stated that the Modified Ashworth Scale is a reliable tool for assessing spasticity in clinical practice. Additionally, it has been emphasized that MAS plays an important role in treatment planning, particularly in neurological rehabilitation processes, for measuring spasticity and monitoring treatment response.

Autonomic Nervous System Assessment:

This system cannot be evaluated directly through physiological tests. With advancements in technology, new methods have been developed, many of which are used in scientific research. The most commonly used method is heart rate variability (HRV) analysis. HRV analysis is based on observing RR waves during rest, and this method will be used in our study using the Elite HRV Corsense device. The values measured by the device are as follows:

RMSSD: Represents the parasympathetic branch of the autonomic nervous system and forms the basis of the HRV score.

LF Power: Reflects the activity in the 0.04-0.15 Hz frequency range and is proportional to sympathetic nervous system activity.

HF Power: Reflects the activity in the 0.15-0.40 Hz frequency range and represents parasympathetic activity. It is highly correlated with time-domain measurements such as PNN50 and RMSSD.

LF/HF Ratio: Represents the ratio of low-frequency power to high-frequency power and is commonly used as a measure of sympathovagal balance, indicating the balance between the opposing branches of the autonomic nervous system.

Average Heart Rate All assessments will be performed by the same expert physiotherapist to ensure standardization.

Treatment Since the acute effect is to be measured, auricular vagus nerve stimulation will be applied once, and pre- and post-intervention evaluations will be conducted.

Auricular Vagus Nerve Stimulation:

Vagus nerve stimulation is a treatment method involving the electrical stimulation of the vagus nerve. Auricular vagus nerve stimulation is a neuromodulation technique performed through the ear, targeting the more accessible part of the vagus nerve. Stimulating the vagus nerve can modulate the interaction between the brain and body and alter neurotransmitter levels. The vagus nerve is superficially located in the ear, particularly in the tragus region, and electrical stimulation applied here activates the nerve. For this purpose, intra-ear electrical stimulation devices are used.

Vagus stimulation will be applied bilaterally through the ear in a transcutaneous manner. taVNS will be performed using the Vagustim portable device. The device is certified, and the certificate will be provided as additional documentation. The stimulation will be applied with a pulse width of 300 microseconds, a frequency of 10 Hz, and in a biphasic manner for 20 minutes. Electrodes will be placed on the concha and tragus parts of the ear, and the current will be increased until the participant feels it.

Statistical Method(s) to be Used:

The sample size was calculated as 14 based on the HF value in the study by Amichai and Katz-Leurer. Using the G*Power 3.1 program, an independent t-test scenario with d: 1.1052191, α: 0.05, and 1-β: 0.95 was selected, and the minimum required sample size was determined to be 14. It is planned to include at least 14 individuals who meet the inclusion criteria, do not meet the exclusion criteria, and volunteer to participate.

The normality of the collected data will be tested using the Kolmogorov-Smirnov and Shapiro-Wilk tests. Parametric statistical methods will be used if the data follow a normal distribution, and non-parametric methods will be used if they do not. Descriptive statistics for continuous variables will be presented as min, max, median, and mean ± standard deviation, while categorical variables will be presented as numbers and percentages.

The data will be analyzed using the SPSS 25.0 software package. Continuous variables will be expressed as mean ± standard deviation, and categorical variables will be expressed as numbers and percentages. Relationships between continuous variables will be examined using Spearman or Pearson correlation analyses, and differences between categorical variables will be examined using the Chi-square test. Additionally, regression models will be constructed to investigate the effects of the variables.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of spastic CP,
* Individuals aged 2-15 years,
* Written informed consent from parents or legal guardians and the willingness of the children to participate in the study,
* Clinically stable children without acute illnesses or comorbidities that could affect autonomic function or spasticity during the study period.

Exclusion Criteria:

* Children with severe intellectual disabilities who cannot understand or respond to the study procedures,
* Children with uncontrolled cardiovascular, respiratory, or autonomic disorders (e.g., arrhythmia, severe asthma),
* Children with devices such as pacemakers or cochlear implants that could be affected by vagus nerve stimulation,
* Children for whom vagus nerve stimulation may interact with antiepileptic drugs or affect seizures,
* Children or parents who cannot comply with the study protocol or cooperate.

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Muscle Spastisity Value | The assessments will be conducted before and immediately after the application of vagus nerve stimulation (VNS).
  The Modified Ashworth Scale (MAS) is a widely used tool to assess spasticity, measuring muscle tone in conditions like cerebral palsy, stroke, and spinal cord injuries. Spasticity causes abnormal muscle contractions and movement limitations. MAS evaluates muscle resistance during joint movements, grading spasticity from 0 (no spasticity) to 4 (joint movement impossible due to high muscle tone). It provides a simple, quick, and reliable method for monitoring spasticity, aiding in treatment planning and rehabilitation. Studies, such as Bohannon and Smith (1987), confirm its reliability in clinical practice, making it valuable for assessing treatment response and intervention needs.
Autonomic Nervous System Activity Value/RMSSD | The assessments will be conducted before and immediately after the application of vagus nerve stimulation (VNS).
  The autonomic nervous system cannot be directly evaluated through physiological tests. However, advancements in technology have introduced methods like heart rate variability (HRV) analysis, widely used in scientific research. HRV analysis measures RR waves during rest and will be employed in this study using the Elite HRV Corsense device. Key parameters include:
  RMSSD: Reflects parasympathetic activity and forms the basis of HRV and and is expressed in milliseconds
Autonomic nervous system activity/ LF Power | The assessments will be conducted before and immediately after the application of vagus nerve stimulation (VNS).
  The autonomic nervous system cannot be directly evaluated through physiological tests. However, advancements in technology have introduced methods like heart rate variability (HRV) analysis, widely used in scientific research. HRV analysis measures RR waves during rest and will be employed in this study using the Elite HRV Corsense device.LF Power: Indicates sympathetic activity (0.04-0.15 Hz range) and t is expressed as the square of milliseconds
Autonomic nervous system activity / HF Power | The assessments will be conducted before and immediately after the application of vagus nerve stimulation (VNS).
  The autonomic nervous system cannot be directly evaluated through physiological tests. However, advancements in technology have introduced methods like heart rate variability (HRV) analysis, widely used in scientific research. HRV analysis measures RR waves during rest and will be employed in this study using the Elite HRV Corsense device.HF Power: Represents parasympathetic activity (0.15-0.40 Hz range) and t is expressed as the square of milliseconds
Autonomic nervous system activity - LF/HF | The assessments will be conducted before and immediately after the application of vagus nerve stimulation (VNS).
  The autonomic nervous system cannot be directly evaluated through physiological tests. However, advancements in technology have introduced methods like heart rate variability (HRV) analysis, widely used in scientific research. HRV analysis measures RR waves during rest and will be employed in this study using the Elite HRV Corsense device.LF/HF Ratio: Measures sympathovagal balance.
Heart Rate | The assessments will be conducted before and immediately after the application of vagus nerve stimulation (VNS).
  HRV analysis measures RR waves during rest and will be employed in this study using the Elite HRV Corsense device.The participants' average heart rate will be recorded in beats per minute (bpm).

SECONDARY OUTCOMES:
Regression Analysis of Gross Motor Function Classification System (GMFCS) Levels | Regression analysis will use post-stimulation data, comparing baseline GMFCS, spasticity, and autonomic activity to assess GMFCS's predictive role in vagus nerve stimulation effectiveness.
  Change from baseline in spasticity, measured using the Modified Ashworth Scale, at 6 weeks post-vagus nerve stimulation. Change in autonomic nervous system activity, evaluated through heart rate variability parameters (RMSSD, LF power, HF power, and LF/HF ratio). The relationship between these changes and participants' baseline Gross Motor Function Classification System (GMFCS) levels will also be analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Mudanya University, Bursa, Bursa, Turkey (Türkiye)